CLINICAL TRIAL: NCT03603106
Title: Assessment of Pharmacokinetics, Pharmacodynamics Profile and Tolerance of P03277 in Healthy Subjects and Patients With Brain Lesions
Brief Title: Pharmacokinetics, Pharmacodynamics Profile and Tolerance of P03277 in Healthy Subjects and Patients With Brain Lesions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Diagnostic
Other Study IDs: GDX-44-003; 2013-004428-12 (EudraCT Number)
Record Dates: First submitted 2018-07-16; First posted 2018-07-27 (Actual); Results first posted 2019-07-12 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers; Brain Lesion
MeSH Terms: interventions — gadopiclenol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Part I: Sequential administration within each group of healthy subjects was established.
  Part II: The administration to patients within the same day was sequential to ensure the well-being of the patients. At least a 1-hour interval between 2 administrations had to be respected.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I (Phase I) (Experimental): In each dose group (0.025, 0.05, 0.075, 0.1, 0.2 and 0.3 mmol/kg), 9 healthy subjects were to be included: 6 subjects received P03277 and 3 subjects received placebo in one single intravenous administration.
  Interventions: Drug: P03277; Drug: Placebo
- Part II (Phase IIA) (Experimental): In each dose group (0.05, 0.075, 0.1 and 0.2 mmol/kg), all 3 patients received one single intravenous administration of P03277.
  Interventions: Drug: P03277

INTERVENTIONS:
Drug: P03277 — Part I: P03277 was administered intravenously with a flow rate ranging from 0.5 to 2 mL/s.
  Part II: P03277 was administered intravenously with a flow rate of 2 mL/s.
  Other Names: Gadopiclenol
Drug: Placebo — Part I: Placebo was administered intravenously with a flow rate ranging from 0.5 to 2 mL/s.
  Part II: Placebo was administered intravenously with a flow rate of 2 mL/s.
  Other Names: NaCl 0.9%
  Arms: Part I (Phase I)

SUMMARY:
The primary objective of this study was to evaluate the safety (clinical and biological) and pharmacokinetics (plasma and urine) profile of P03277 following single administration at ascending dose levels in healthy subjects.

DETAILED DESCRIPTION:
This single-center, single ascending dose, phase I/IIa study was divided into 2 parts, involving both healthy subjects and patients with brain lesions:

* Study Part I included healthy subjects: double-blind, randomized, placebo control;
* Study Part II included patients with brain lesions: open-label.

In Part I, the following 6 dosing groups were investigated:

* Group 1: 0.025 mmol/kg
* Group 2: 0.05 mmol/kg
* Group 3: 0.075 mmol/kg
* Group 4: 0.1 mmol/kg
* Group 5: 0.2 mmol/kg
* Group 6: 0.3 mmol/kg

Healthy subjects were included and were then administered with P03277 or placebo and were to undergo MRI examination according to the randomization scheme.

In Part II, the following 4 doses groups were investigated:

* Group 7: 0.05 mmol/kg
* Group 8: 0.075 mmol/kg
* Group 9: 0.1 mmol/kg
* Group 10: 0.2 mmol/kg

Patients with brain lesions were included and were then administered with P03277 and underwent MRI examination.

ELIGIBILITY:
Inclusion Criteria:

* Part I: Subjects between 18 and 45 years old (inclusive), with a body mass index (BMI) of 18 to 30 kg/m² (exclusive) and in a good health.
* Part II: Patients 18 years old and older and having at least one brain lesion with a disruption of the blood brain barrier (BBB) and/or with abnormal vascularity in the brain. This/these lesion(s) must have been detected by previous imaging evaluation (Computed Tomography or MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2015-04-17 (Actual); Study Completion 2015-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Haazen, MD, Principal Investigator — SGS Clinical Pharmacology Unit
Locations (1):
- Clinical Pharmacology unit, SGS Life Science Services, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hao J, Bourrinet P, Desche P. Assessment of Pharmacokinetic, Pharmacodynamic Profile, and Tolerance of Gadopiclenol, A New High Relaxivity GBCA, in Healthy Subjects and Patients With Brain Lesions (Phase I/IIa Study). Invest Radiol. 2019 Jul;54(7):396-402. doi: 10.1097/RLI.0000000000000556. PMID 30870257

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For part I, all patients who were not randomized were screening failures. For part II, all patients who were not allocated to a dose of P03277 were screening failures.
Groups:
- Part I (Phase I) P03277 0.025 mmol/kg: 6 subjects received P03277 in one single administration. P03277 was administered intravenously at 0.025 mmol/kg with a flow rate ranging from 0.5 to 2 mL/s.
- Part I (Phase I) P03277 0.05 mmol/kg: 6 subjects received P03277 in one single administration. P03277 was administered intravenously at 0.05 mmol/kg with a flow rate ranging from 0.5 to 2 mL/s.
- Part I (Phase I) P03277 0.075 mmol/kg: 6 subjects received P03277 in one single administration. P03277 was administered intravenously at 0.075 mmol/kg with a flow rate ranging from 0.5 to 2 mL/s.
- Part I (Phase I) P03277 0.1 mmol/kg: 6 subjects received P03277 in one single administration. P03277 was administered intravenously at 0.1 mmol/kg with a flow rate ranging from 0.5 to 2 mL/s.
- Part I (Phase I) P03277 0.2 mmol/kg: 6 subjects received P03277 in one single administration. P03277 was administered intravenously at 0.2 mmol/kg with a flow rate ranging from 0.5 to 2 mL/s.
- Part I (Phase I) P03277 0.3 mmol/kg: 6 subjects received P03277 in one single administration. P03277 was administered intravenously at 0.3 mmol/kg with a flow rate ranging from 0.5 to 2 mL/s.
- Part I (Phase I) Placebo: 3 healthy subjects per dose group received placebo in one single administration.
  Placebo was administered intravenously with a flow rate ranging from 0.5 to 2 mL/s.
- Part II (Phase IIA) P03277 0.05 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.05 mmol/kg with a flow rate of 2 mL/s.
- Part II (Phase IIA) P03277 0.075 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.075 mmol/kg with a flow rate of 2 mL/s.
- Part II (Phase IIA) P03277 0.1 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.1 mmol/kg with a flow rate of 2 mL/s.
- Part II (Phase IIA) P03277 0.2 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.2 mmol/kg with a flow rate of 2 mL/s.
Period: Overall Study
Arm/Group | Part I (Phase I) P03277 0.025 mmol/kg | Part I (Phase I) P03277 0.05 mmol/kg | Part I (Phase I) P03277 0.075 mmol/kg | Part I (Phase I) P03277 0.1 mmol/kg | Part I (Phase I) P03277 0.2 mmol/kg | Part I (Phase I) P03277 0.3 mmol/kg | Part I (Phase I) Placebo | Part II (Phase IIA) P03277 0.05 mmol/kg | Part II (Phase IIA) P03277 0.075 mmol/kg | Part II (Phase IIA) P03277 0.1 mmol/kg | Part II (Phase IIA) P03277 0.2 mmol/kg
Started | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 3 | 3 | 3 | 3
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received one injection of product (placebo or P03277 for Part I, P03277 for Part II).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I (Phase I) P03277 0.025 mmol/kg | Part I (Phase I) P03277 0.05 mmol/kg | Part I (Phase I) P03277 0.075 mmol/kg | Part I (Phase I) P03277 0.1 mmol/kg | Part I (Phase I) P03277 0.2 mmol/kg | Part I (Phase I) P03277 0.3 mmol/kg | Part I (Phase I) Placebo | Part II (Phase IIA) P03277 0.05 mmol/kg | Part II (Phase IIA) P03277 0.075 mmol/kg | Part II (Phase IIA) P03277 0.1 mmol/kg | Part II (Phase IIA) P03277 0.2 mmol/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 3 | 3 | 3 | 3 | 66
Age, Continuous [Median (Full Range); unit: years] | 26.0 [22 to 30] | 25.5 [21 to 37] | 27.5 [23 to 40] | 25.5 [23 to 41] | 23.0 [18 to 36] | 33.5 [23 to 42] | 26.5 [19 to 43] | 40.0 [37 to 50] | 56.0 [25 to 57] | 56.0 [53 to 61] | 53.0 [50 to 58] | 28.0 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 3 | 3 | 3 | 8 | 1 | 2 | 1 | 1 | 32
  Male | 3 | 2 | 3 | 3 | 3 | 3 | 10 | 2 | 1 | 2 | 2 | 34
Weight [Median (Full Range); unit: kg] | 81.65 [52.2 to 87.4] | 71.60 [54.0 to 83.6] | 65.00 [56.4 to 93.0] | 72.50 [62.0 to 99.2] | 69.30 [68.2 to 87.6] | 72.50 [61.6 to 88.6] | 67.90 [56.8 to 89.4] | 87.20 [85.8 to 89.0] | 80.40 [71.2 to 87.4] | 87.20 [82.4 to 102.8] | 85.80 [79.4 to 101.6] | 72.85 [52.2 to 102.8]

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter Cmax
Description: Cmax = maximum concentration measured. Blood samples were taken to assess the P03277 concentration.
Time Frame: From baseline (30 minutes before injection) to 24 hours post-injection
Population: In part I, one patient from the "0.025 mmol/kg" group was excluded from the pharmacokinetics analysis (incorrect volume of P03277 injected).
  In part II, one patient from the "0.1 mmol/kg" group was excluded from the pharmacokinetics analysis (incorrect route of administration, high probability of extravasation).
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Part II (Phase IIA) 0.05 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.05 mmol/kg with a flow rate of 2 mL/s.
- Part II (Phase IIA) 0.075 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.075 mmol/kg with a flow rate of 2 mL/s.
- Part II (Phase IIA) 0.1 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.1 mmol/kg with a flow rate of 2 mL/s.
- Part II (Phase IIA) 0.2 mmol/kg: 3 patients received one single administration of P03277. P03277 was administered intravenously at 0.2 mmol/kg with a flow rate of 2 mL/s.
Arm/Group | Part I (Phase I) P03277 0.025 mmol/kg | Part I (Phase I) P03277 0.05 mmol/kg | Part I (Phase I) P03277 0.075 mmol/kg | Part I (Phase I) P03277 0.1 mmol/kg | Part I (Phase I) P03277 0.2 mmol/kg | Part I (Phase I) P03277 0.3 mmol/kg | Part II (Phase IIA) 0.05 mmol/kg | Part II (Phase IIA) 0.075 mmol/kg | Part II (Phase IIA) 0.1 mmol/kg | Part II (Phase IIA) 0.2 mmol/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 2 | 3
µg/mL | 248.7 (54.5) | 524.5 (69.9) | 698.7 (378.9) | 992.0 (233.1) | 2097.6 (572.3) | 3916.4 (1114.8) | 370.8 (117.6) | 618.2 (439.7) | 701.6 (48.5) | 1434.9 (651.5)

2. Primary Outcome: PK Parameter T1/2
Description: T1/2 = terminal elimination half-life of the compound. Blood samples were taken to assess the P03277 concentration.
Time Frame: From baseline (30 minutes before injection) to 24 hours post-injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Part I (Phase I) P03277 0.025 mmol/kg; Part I (Phase I) P03277 0.05 mmol/kg; Part I (Phase I) P03277 0.075 mmol/kg; Part I (Phase I) P03277 0.1 mmol/kg; Part I (Phase I) P03277 0.2 mmol/kg; Part I (Phase I) P03277 0.3 mmol/kg: 6 subjects received P03277 in one single administration. P03277 was administered intravenously with a flow rate ranging from 0.5 to 2 mL/s.
- Part II (Phase IIA) 0.05 mmol/kg; Part II (Phase IIA) 0.075 mmol/kg; Part II (Phase IIA) 0.1 mmol/kg; Part II (Phase IIA) 0.2 mmol/kg: In each dose group, all 3 patients received one single administration of P03277.
  P03277 was administered intravenously with a flow rate of 2 mL/s.
Arm/Group | Part I (Phase I) P03277 0.025 mmol/kg | Part I (Phase I) P03277 0.05 mmol/kg | Part I (Phase I) P03277 0.075 mmol/kg | Part I (Phase I) P03277 0.1 mmol/kg | Part I (Phase I) P03277 0.2 mmol/kg | Part I (Phase I) P03277 0.3 mmol/kg | Part II (Phase IIA) 0.05 mmol/kg | Part II (Phase IIA) 0.075 mmol/kg | Part II (Phase IIA) 0.1 mmol/kg | Part II (Phase IIA) 0.2 mmol/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 2 | 3
hours | 1.65 (0.43) | 1.50 (0.22) | 1.58 (0.30) | 1.73 (0.26) | 1.82 (0.35) | 2.09 (0.15) | 1.90 (0.04) | 2.04 (0.06) | 1.79 (0.17) | 1.94 (0.06)

3. Primary Outcome: PK Parameter Cl
Description: Cl = total clearance. Blood samples were taken to assess the P03277 concentration.
Time Frame: From baseline (30 minutes before injection) to 24 hours post-injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Part I (Phase I) P03277 0.025 mmol/kg | Part I (Phase I) P03277 0.05 mmol/kg | Part I (Phase I) P03277 0.075 mmol/kg | Part I (Phase I) P03277 0.1 mmol/kg | Part I (Phase I) P03277 0.2 mmol/kg | Part I (Phase I) P03277 0.3 mmol/kg | Part II (Phase IIA) 0.05 mmol/kg | Part II (Phase IIA) 0.075 mmol/kg | Part II (Phase IIA) 0.1 mmol/kg | Part II (Phase IIA) 0.2 mmol/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 2 | 3
mL/min | 91.7 (8.5) | 100.1 (9.5) | 106.4 (20.7) | 96.1 (11.8) | 101.3 (10.9) | 102.2 (19.0) | 105.3 (13.5) | 106.5 (15.7) | 108.6 (5) | 109.9 (18.2)

4. Primary Outcome: PK Parameter Vd
Description: Vd = volume of distribution. Blood samples were taken to assess the P03277 concentration.
Time Frame: From baseline (30 minutes before injection) to 24 hours post-injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Part I (Phase I) P03277 0.025 mmol/kg | Part I (Phase I) P03277 0.05 mmol/kg | Part I (Phase I) P03277 0.075 mmol/kg | Part I (Phase I) P03277 0.1 mmol/kg | Part I (Phase I) P03277 0.2 mmol/kg | Part I (Phase I) P03277 0.3 mmol/kg | Part II (Phase IIA) 0.05 mmol/kg | Part II (Phase IIA) 0.075 mmol/kg | Part II (Phase IIA) 0.1 mmol/kg | Part II (Phase IIA) 0.2 mmol/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 2 | 3
mL | 13203 (4122) | 12945 (1692) | 14312 (2742) | 14351 (2645) | 15922 (3224) | 18487 (3575) | 17320 (1942) | 18796 (2478) | 16823 (804) | 18355 (2522)

ADVERSE EVENTS:
Time Frame: For Part I: adverse events were collected from subjects' enrollment until 7 days after the product (P03277 or placebo) administration. For Part II: adverse events were collected from patients' enrollment until 1 day after P03277 administration.
Description: All adverse events occuring pre- and post-injection are reported below.
Arm/Group | Part I (Phase I) P03277 0.025 mmol/kg | Part I (Phase I) P03277 0.05 mmol/kg | Part I (Phase I) P03277 0.075 mmol/kg | Part I (Phase I) P03277 0.1 mmol/kg | Part I (Phase I) P03277 0.2 mmol/kg | Part I (Phase I) P03277 0.3 mmol/kg | Part I (Phase I) Placebo | Part II (Phase IIA) P03277 0.05 mmol/kg | Part II (Phase IIA) P03277 0.075 mmol/kg | Part II (Phase IIA) P03277 0.1 mmol/kg | Part II (Phase IIA) P03277 0.2 mmol/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/18 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/18 | 0/3 | 1/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 2/6 | 4/6 | 5/6 | 3/6 | 11/18 | 1/3 | 1/3 | 1/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I (Phase I) P03277 0.025 mmol/kg (N=6) | Part I (Phase I) P03277 0.05 mmol/kg (N=6) | Part I (Phase I) P03277 0.075 mmol/kg (N=6) | Part I (Phase I) P03277 0.1 mmol/kg (N=6) | Part I (Phase I) P03277 0.2 mmol/kg (N=6) | Part I (Phase I) P03277 0.3 mmol/kg (N=6) | Part I (Phase I) Placebo (N=18) | Part II (Phase IIA) P03277 0.05 mmol/kg (N=3) | Part II (Phase IIA) P03277 0.075 mmol/kg (N=3) | Part II (Phase IIA) P03277 0.1 mmol/kg (N=3) | Part II (Phase IIA) P03277 0.2 mmol/kg (N=3)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I (Phase I) P03277 0.025 mmol/kg (N=6) | Part I (Phase I) P03277 0.05 mmol/kg (N=6) | Part I (Phase I) P03277 0.075 mmol/kg (N=6) | Part I (Phase I) P03277 0.1 mmol/kg (N=6) | Part I (Phase I) P03277 0.2 mmol/kg (N=6) | Part I (Phase I) P03277 0.3 mmol/kg (N=6) | Part I (Phase I) Placebo (N=18) | Part II (Phase IIA) P03277 0.05 mmol/kg (N=3) | Part II (Phase IIA) P03277 0.075 mmol/kg (N=3) | Part II (Phase IIA) P03277 0.1 mmol/kg (N=3) | Part II (Phase IIA) P03277 0.2 mmol/kg (N=3)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site dermatitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site coldness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other